CLINICAL TRIAL: NCT00612508
Title: The Effects of Oral vs. Intravaginal Hormonal Contraception on Vaginal Health
Brief Title: Hormonal Contraception and Vaginal Health
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Oregon Health and Science University (Other)
Collaborators: Oregon Clinical and Translational Research Institute (Other)
Responsible Party: Principal Investigator, Jeffrey Jensen, MD MPH, Oregon Health and Science University
Allocation: Randomized | Model: Parallel | Masking: None
Other Study IDs: OHSU RES 2017
Record Dates: First submitted 2008-01-29; First posted 2008-02-11 (Estimated); Results first posted 2012-11-08 (Estimated); Last update posted 2012-11-08 (Estimated); Status verified 2012-10

CONDITIONS: Contraceptive Usage; Vaginal Epithelial Disruption
Keywords: contraception; NuvaRing; Desogen; vaginal biopsy
MeSH Terms: conditions — Contraception Behavior | interventions — Desogestrel; Ethinyl Estradiol; NuvaRing; etonogestrel

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Desogen (Active Comparator): Drug: ethinyl estradiol and desogestrel
  1 tablet every day; each tablet contains 0.15mg desogestrel and 0.03mg ethinyl estradiol; secen inactive pills every 28 days.
  Subjects receive baseline vaginal biopsy, followed by treatment with the OC for six cycles and repeat biopsy at 3 and after 6 cycles
  Interventions: Drug: Desogen (ethinyl estradiol and desogestrel)
- NuvaRing (Active Comparator): Intravaginal Contraception
  ethinyl estradiol (0.15 mg/d) and etonogestrel (0.12 mg/d) Place the ring in the vagina for 3 weeks, remove for one week. Repeat with new Ring
  Subjects had baseline vaginal biopsy followed by 6 cycles of ring use and repeat biopsy at 3 and after 6 cycles
  Interventions: Drug: NuvaRing (ethinyl estradiol and etonogestrel)

INTERVENTIONS:
Drug: Desogen (ethinyl estradiol and desogestrel) — 1 tablet every day; each tablet contains 0.15mg desogestrel and 0.03mg ethinyl estradiol
  Other Names: Desogen®
  Arms: Desogen
Drug: NuvaRing (ethinyl estradiol and etonogestrel) — Place the ring in the vagina for 3 weeks, remove for one week. Repeat with new Ring
  Other Names: NuvaRing®
  Arms: NuvaRing

SUMMARY:
The purpose of this study is to help determine if the route by which women receive hormonal contraception causes different changes to occur in the lining of the vagina. The investigators plan to compare an oral route (taking birth control pills) with a vaginal route (using a vaginal ring).

DETAILED DESCRIPTION:
The investigators intend to conduct a prospective, randomized study at Oregon Health and Science University. This study will be conducted over six 28-day cycles. Subjects enrolled in the study will undergo baseline vaginal biopsy and then be randomized to receive either intravaginal ethinyl estradiol and etonogestrel (NuvaRing®) or oral ethinyl estradiol and desogestrel (Desogen®). Repeat vaginal biopsies will be obtained after three and six months of exposure to either oral or intravaginal hormonal contraception. These will be analyzed to measure the thickness of the vaginal epithelium and to quantify the presence of Langerhans cell, macrophages, T-lymphocytes and dendritic cells.

ELIGIBILITY:
Inclusion Criteria:

* Female
* 18-35 years
* In general good health
* With regular menses (every 28-32 days)
* Seeking contraception and willing to use a hormonal method for at least 6 months

Exclusion Criteria:

* Current or recent (within the past 8 weeks) vaginitis or pelvic inflammatory disease
* History of recurrent vaginitis (> 2 episodes in one year, any type)
* Pregnancy
* Recent use of hormonal contraceptives
* Depot medroxyprogesterone: 6 months
* Progestin implants: 3 months
* Oral contraceptives: 3 months
* Hormone impregnated IUD: 3 months
* Contraindications to use of oral contraceptive pills or vaginal ring
* History of deep vein thrombosis
* Known coagulopathy or thrombophilia
* Unexplained vaginal bleeding
* Uncontrolled hypertension
* Diabetes with vascular changes
* Present or history of hepatic disease or liver tumors
* Migraines with neurologic changes
* Myocardial infection
* Pulmonary embolus
* Stroke
* Breast cancer
* Hypersensitivity or allergy to hormonal contraception
* Heavy Smoking ( ≥ 15 cigarettes per day)

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 14 (Actual)
Dates: Start 2007-05; Primary Completion 2008-05 (Actual); Study Completion 2008-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey T Jensen, MD., MPH, Principal Investigator — Oregon Health and Science University
Locations (1):
- Oregon Health and Science University, Portland, Oregon, United States

REFERENCES:
- See also: (Women's Health Research Unit website) — http://www.ohsuwomenshealth.com/research/index.html

RESULTS

PARTICIPANT FLOW:
Groups:
- Desogen: oral contraceptive
- NuvaRing: intravaginal contraception
Period: Overall Study
Arm/Group | Desogen | NuvaRing
Started | 7 | 7
Completed | 4 (5 desogen users returned for the 84 day biopsy) | 3 (6 nuvaring users returned for the 84 day biopsy)
Not Completed | 3 | 4
Not completed — Withdrawal by Subject | 3 | 4

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Desogen | NuvaRing | Total
Number analyzed (Participants) | 7 | 7 | 14
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 7 | 7 | 14
  >=65 years | 0 | 0 | 0
Age Continuous [Mean (Standard Deviation); unit: years] | 28 (4) | 24 (3.4) | 25.8 (4.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 7 | 14
  Male | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 7 | 7 | 14

OUTCOME MEASURES:

1. Primary Outcome: Thickness of the Vaginal Epithelium (in mm)With Means and Standard Deviations Reported.
Description: Histologic evalation of vaginal sections was performed to measured and record the absolute thickness of the vaginal epithelium. Baseline findings were compared to biopsies after three and six cycles of treatment. Mean values were compared using T-test for paired data for baseline and 84 days, and baseline and 168 days
Time Frame: baseline, 84 days, 168 days
Population: A total of 14 subjects (7 R, 7 P) were randomized and had an initial biopsy; 11 (6 R, 5 P) returned for a biopsy at 3rd cycle (84 days), and 6 (3 R, 4 P) 6th cycle (168 days).
  The analysis used a paired T test comparing the baseline mean to the mean as the end of the 3rd cylce (e.g. 84 days) and the 6th cycle (168 days)
Measure: Mean (Standard Deviation); unit: mm
Groups:
- Desogen: oral contraceptive = P (pill)
- NuvaRing: intravaginal contraception = R (ring)
Arm/Group | Desogen | NuvaRing
Number analyzed (Participants) | 5 | 6
mm
  mean difference at 84 days | 0.01 (0.06) | -0.005 (0.048)
  mean difference at 168 days | -0.02 (0.09) | .007 (0.028)

2. Secondary Outcome: Adverse Events
Description: Self-reported treatment-related and serious adverse events
Time Frame: over 168 days
Population: All subjects that were enrolled were assessed for adverse events at each study visit. Measure is number of participants with event
Measure: Number; unit: participants
Groups:
- Oral Contraceptive: Desogen (ethinyl estradiol & desogestrel) = P (pill)
- Intravaginal Ring Contraceptive: nuvaring (ethinyl estradiol & desogestrel) = R (ring)
Arm/Group | Oral Contraceptive | Intravaginal Ring Contraceptive
Number analyzed (Participants) | 7 | 7
participants | 1 | 0

ADVERSE EVENTS:
Time Frame: Every 6 months
Arm/Group | Desogen | NuvaRing
Serious Adverse Events (participants affected / at risk) | 0/7 | 0/7
Other Adverse Events (participants affected / at risk) | 1/7 | 0/7
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Desogen (N=7) | NuvaRing (N=7)
Bleeding from vagina (Reproductive system and breast disorders) | 1 (1) | 0 (0) — Minor bleeding and pain associated with biopsy

LIMITATIONS AND CAVEATS:
Did not fully recruit; small number of subject

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No